CLINICAL TRIAL: NCT02892591
Title: A Double-Blind, Placebo-Controlled Crossover Study Comparing the Analgesic Efficacy of Cannabis Versus Oxycodone
Brief Title: Cannabis Versus Oxycodone for Pain Relief
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-1909
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Back Pain; Neck Pain
MeSH Terms: conditions — Back Pain; Neck Pain | interventions — nabiximols; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cannabis (Experimental): Medium dose THC, single administration, vaporized
  Interventions: Drug: Cannabis; Drug: Placebo for Oxycodone
- Oxycodone (Active Comparator): 5-10 mg oxycodone hydrochloride, single administration, oral
  Interventions: Drug: Oxycodone; Drug: Placebo for Cannabis
- Placebo (Placebo Comparator): No active study drug
  Interventions: Drug: Placebo for Cannabis; Drug: Placebo for Oxycodone

INTERVENTIONS:
Drug: Cannabis — vaporized plant material
  Other Names: marijuana
  Arms: Cannabis
Drug: Oxycodone — oral capsule
  Arms: Oxycodone
Drug: Placebo for Cannabis — vaporized placebo plant material
  Arms: Oxycodone; Placebo
Drug: Placebo for Oxycodone — oral placebo capsule
  Arms: Cannabis; Placebo

SUMMARY:
This study investigates the ability of cannabis to reduce chronic back and neck pain and to reduce sensitivity to an acute painful stimulus. Cannabis will be compared to both oxycodone and a placebo.

DETAILED DESCRIPTION:
This study investigates the ability of cannabis to reduce chronic back and neck pain and to reduce sensitivity to an acute painful stimulus. Cannabis will be compared to both oxycodone and a placebo.

Some inclusion/exclusion criteria are purposely omitted at this time to preserve scientific integrity. They will be included after the trial is complete.

ELIGIBILITY:
Overall Inclusion Criteria:

* Previous smoked or vaporized cannabis exposure
* Age ≥21 years

Overall Exclusion Criteria:

* Current substance use disorder
* Current alcohol use disorder
* Past cannabis abuse/dependence
* Current use of amphetamine/methamphetamine, barbiturates, benzodiazepines, cocaine, phencyclidine (PCP), MDMA (ecstasy)
* Prior adverse reaction to cannabis exposure (paranoia, anxiety, etc.)
* Allergy to or prior adverse reaction to oxycodone
* Any condition contraindicative to opioid use (e.g. paralytic ileus)
* History or diagnosis of schizophrenia or bipolar disorder
* Current severe depression
* Uncontrolled hypertension (>139/89)
* Known cardiovascular disease
* Known immune system disorder
* Chronic pulmonary disease (e.g., bronchitis, asthma, COPD, or emphysema)
* History of seizure disorder
* Diagnosed inflammatory disease (e.g. Rheumatoid Arthritis (RA))
* Clinically significant abnormal values on CBC/CMP/EKG tests
* Cognitive disability that interferes with ability to provide consent or understand study procedures
* Inability to refrain from using tobacco for at least 4 hours
* Pregnant females
* Lactating females

Additional Exclusion Criteria for SPINE PATIENTS

* Current regular use of a long acting opioid (e.g. OxyContin, MS Contin, other extended release formulas)
* Current high-dose use of immediate release opioid
* Current high-dose use of nerve-targeted medication
* Other diagnosed chronic pain syndromes of greater severity than spine condition (e.g. knee pain )
* Diagnosed Fibromyalgia
* Neuropathy not associated with spine condition (e.g. diabetic neuropathy)

Additional Exclusion Criteria for HEALTHY CONTROLS

* Current acute pain
* Current chronic pain condition (e.g. fibromyalgia, neuropathy)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Pain Numeric Rating Scale (NRS) score (Spine Patients) | 3 hours
Pain Threshold (kPa) (Healthy Controls) | 3 hours

SECONDARY OUTCOMES:
Patient Global Impression of Change score | 3 hours
Drug effect rating | 3 hours
Psychoactive effect rating | 3 hours
Mood rating | 3 hours
Symbol Digit Modalities Test (SDMT) | 3 hours
Hopkins Verbal Learning Test Revised (HVLT) | 3 hours
Standardized Field Sobriety Test | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Emily Lindley, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States